CLINICAL TRIAL: NCT00607776
Title: Artificial Tears Study in Mild to Moderate Dry Eye Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Lynn Lasswell, O.D., Director, Eye Care Clinical Research, AMO, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEGT-104-9582
Record Dates: First submitted 2007-12-19; First posted 2008-02-06 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
Keywords: dry, eyes; Amelioration of dry eye symptoms
MeSH Terms: conditions — Dry Eye Syndromes; Xerophthalmia | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Systane
  Interventions: Drug: Systane
- 2 (Experimental): Blink tears
  Interventions: Drug: (9587X) Blink Tears, classified as an OTC Drug with the active ingredient being plyethylene glycol 400

INTERVENTIONS:
Drug: (9587X) Blink Tears, classified as an OTC Drug with the active ingredient being plyethylene glycol 400 — Drops
  Arms: 2
Drug: Systane — Drops
  Arms: 1

SUMMARY:
The mean change in the subjective comfort score from baseline of the test group is at least 2.0 units less than that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate dry eye
* over 18

Exclusion Criteria:

* No concurrent ocular disease or meds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Subjective ocular comfort | 1 Month

SECONDARY OUTCOMES:
Vision quality | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, M.D., Principal Investigator — Ophthalmic Consultants of Long Island